CLINICAL TRIAL: NCT01605175
Title: Predictors of Tissue Healing in Inflammatory Bowel Disease Patients Treated With Anti-TNF
Brief Title: Predictors of Mucosal Healing in Inflammatory Bowel Disease (IBD) Patients Treated With Anti-TNF
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Collaborators: University of Athens (Other); Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Nikos Viazis, principal investigator - director gastrenterologist, Evangelismos Hospital
Other Study IDs: nviazis
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Predictors Mucosal Healing
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Bowel mucosal tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to prospectively identify, at diagnosis of the disease, factors predictive of mucosal healing in patients with inflammatory bowel disease treated with anti-TNF.

DETAILED DESCRIPTION:
Crohn's disease and ulcerative colitis (UC) are both chronic idiopathic inflammatory conditions of the gastrointestinal tract that result in a considerably decreased quality of life. Long term experience with standard therapies for inflammatory bowel disease patients up to the late 1990s demonstrated diverse limitations. Corticosteroids have good short term efficacy, but are not suitable for maintaining remission, while treatment with immunomodulators are associated with an important risk of side effects. The introduction of monoclonal antibody to tumor necrosis factor a (TNFa) therapy has offered new treatment options originally in patients with Crohn's disease and more recently in those with ulcerative colitis as well. Several clinicians based on the results of clinical trials, now advocate the early use of intensive therapy (immunosuppressants and/or biologics) to maintain a good quality of life from the first flare up and prevent any irreversible consequence of the disease.

Meanwhile, the assessment of tissue healing has become of paramount importance in patients treated for inflammatory bowel disease. Simple clinical assessment does not reflect real activity and inflammation at the tissue level. Moreover, cumulative tissue damage generated by the persisting tissue inflammation leads to non reversible anatomic and functional consequences. Therefore, in order to evaluate both the natural history and impact of treatment in inflammatory bowel disease standardized assessment of tissue healing must be available. Endoscopic and histological healing has been shown to be associated with a reduced risk of recurrence of the disease, in addition to reduced hospitalization and surgery. Furthermore, in patients treated with costly and highly immunosuppressive TNF-a antagonists, achievement of an objective treatment response is essential. Consequently, endoscopic healing should be regarded as the primary approach in the treatment of inflammatory bowel disease.

Although several clinical trials have identified, at diagnosis, factors predictive of a subsequent disabling course of the disease, therefore identifying patients that would mostly benefit from early aggressive therapy with anti-TNF, factors predictive of mucosal healing have not yet been identified.

Endoscopy (ileocolonoscopy) will be performed at baseline (i.e. before anti-TNF administration) for all patients included in the study. The outcome of anti-TNF therapy will be evaluated by two follow up endoscopies, at 3 months and at 12 months after the start of therapy. At the same time periods the disease activity will be documented as well.

For Crohn's disease patients, the simplified endoscopic severity index will be recorded (SES-CD), table 1. According to current guidelines, mucosal healing will be defined as an SES-CD of lower than 5 points. For all CD patients, the CD activity index (CDAI) will also be determined.

For ulcerative colitis, the Mayo endoscopic subscore will be recorded (0: normal mucosa, 1: faded vascular pattern, mild friability, 2: loss of vascular pattern, erosions, friability, 3: ulcers of spontaneous bleeding). According to recent recommendation of the Food and Drug Administration, mucosal healing will be defined as a Mayo score of 0. Disease activity will be graded according to the Clinical Activity Index (Lichtiger's CAI), with a highest possible score of 21. For all ulcerative colitis patients the Montreal classification of the extent of the disease will also be assessed.

Laboratory data on blood hemoglobin, hematocrit, white blood cells, plasma or serum albumin and C-reactive protein (CRP) will be collected for all patients at baseline. Use of concurrent medication will be recorded, especially the dosage data of corticosteroids and those of other immunosuppressant medications.

Infliximab will be administered at 5 mg/Kg body weight at 0, 2 and 6 weeks and thereafter, every 2 months for the follow up period of 1 year. Adalimumab will be administered at a dose of 160mg at week 0, 80 mg at week 2, 40 mg at week 4 and 40 mg every other week thereafter.

The primary goal of this study is to identify predictors, at baseline, for mucosal healing in patients with ulcerative colitis or Crohn's disease that will receive infliximab or adalimumab for control of their disease. For this reason at the end of the follow up period (12 months), the following variables will be tested by univariate analysis:

Patient characteristics at baseline

* age
* gender
* age at onset of disease
* duration of disease
* concomitant corticosteroid use at start of anti_TNF therapy
* concomitant immunosuppressant use at start of anti-TNF therapy
* Blood hemoglobin
* Hematocrit
* White blood cells
* Serum albumin
* C-reactive protein
* Fecal calprotectin level
* CDAI at baseline for CD patients
* Lichtiger score at baseline for UC patients
* Previous major abdominal surgery
* Tobacco use
* Indication for anti-TNF therapy in CD patients (luminal CD, luminal and fistulizing CD, luminal CD with extra-intestinal manifestations)
* Location of disease for CD patients (ileitis, colitis, ileocolitis)
* Location of disease for UC patients (Montreal classification)
* Prior appendectomy

In addition, immunological markers with predictive value for mucosal healing at 1 year will be sought at the intestinal as well the systemic level. Investigators will test these markers both at baseline but also at week 12. In this way, investigators will try to identify pre-treatment predictors of mucosal healing but also early predictors of response to anti-TNF agents.

For the determination of mucosal markers, at endoscopy investigators will collect 2 biopsy samples in RNA-later. These samples will be stored at -80 C, and used for the quantitative messenger ribonucleic acid (mRNA) expression of various immunological markers, mainly cytokines and their receptors, adhesion molecules and other inflammatory proteins by real-time polymerase chain reaction (RT-PCR). A third biopsy specimen will be immersed in formalin and maintained for protein expression studies by immunohistochemistry. Biopsies will be collected both from overtly inflamed and normal-looking mucosa and from various locations when feasible.

For the determination of systemic markers, blood will be collected from the patients and serum separated and stored at -26 C. These samples will be used for the measurement of soluble inflammatory markers that may demonstrate predictive value for the achievement of mucosal healing. Inflammatory markers may be measured by Multiplex assays of by individual ELISAs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Crohn luminal ileitis, colitis or ileocolitis necessitating therapy with anti-TNF, according to the physician's judgment, based on the current European Crohn's and Colitis Organisation (ECCO) guidelines.
* Patients with corticosteroid resistant or corticosteroid dependent ulcerative colitis, necessitating therapy with anti-TNF, according to the physician's judgment, based on the current ECCO guidelines.

Exclusion Criteria:

* Patients with isolated fistulizing or stricturing or upper gastrointestinal Crohn disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with anti-TNF in a tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Endoscopical and histological mucosal healing | 12 weeks

SECONDARY OUTCOMES:
Endoscopical and histological mucosal healing | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Director, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Greece